CLINICAL TRIAL: NCT01055847
Title: A Blinded, Multicenter, Randomized, Placebo-Controlled Trial With Aztreonam for Inhalation (AI) in Cystic Fibrosis Patient With Lung Disease Due to P. Aeruginosa Infection
Brief Title: Aztreonam for Inhalation (AI) in Patients With Cystic Fibrosis & P. Aeruginosa Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Salus Pharma, Inc. (Industry)
Responsible Party: A. Bruce Montgomery, Sr. VP Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-AI-003
Record Dates: First submitted 2010-01-23; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Cystic Fibrosis; CF; Lung Infection; Pseudomonas Aeruginosa
Keywords: cystic fibrosis; CF; aztreonam; lung infection; Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Aztreonam; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AI 75 mg (Experimental): Aztreonam for Inhalation 75 mg twice daily
  Interventions: Drug: Aztreonam for Inhalation (AI)
- AI 225 mg (Experimental): Aztreonam for Inhalation 225 mg twice daily
  Interventions: Drug: Aztreonam for Inhalation (AI)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aztreonam for Inhalation (AI) — Aztreonam for Inhalation
  Other Names: AI
  Arms: AI 225 mg; AI 75 mg
Drug: Placebo — Saline Placebo
  Arms: Placebo

SUMMARY:
This is multicenter placebo-controlled study evaluating the safety and efficacy of AI at two dosage levels compared to placebo in CF patients with P. aeruginosa lung infection.

DETAILED DESCRIPTION:
This is multicenter placebo-controlled study evaluating the safety and efficacy of a 14-day treatment of AI at two dosage levels as compared to placebo, given twice daily, in CF patients with P. aeruginosa lung infection, delivered by the eFlow investigational nebulizer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to the performance of any study related procedures.
* 13 years of age and above.
* Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test (QPIT) or homozygosity for ΔF508 genetic mutation or heterozygosity for two well characterized mutations.
* Ability to perform pulmonary function tests.
* FEV1 ≥ 40% predicted at Visit 1 (Screening).
* SaO2 ≥ 90% at Visit 1 (Screening).
* P. aeruginosa present in sputum at Visit 1 (Screening).
* Ability to expectorate sputum on a daily basis.

Exclusion Criteria:

* Administration of any antibiotic with antipseudomonal activity by any route within 56 days prior to Visit 1 (Screening).
* Administration of any investigational drug or device within 28 days of Visit 1 (Screening) and within 6 half-lives of the investigational drug.
* Oral corticosteroids in doses exceeding 10 mg per day or 20 mg every other day.
* History of sputum culture or throat swab culture yielding B. cepacia in the previous two years.
* Current daily continuous oxygen supplementation or requirement for more than 2 L/min at night.
* Known local or systemic hypersensitivity to monobactam antibiotics.
* Changes in antimicrobial, bronchodilator, anti-inflammatory or corticosteroid medications within 7 days prior to Visit 1 (Screening).
* Changes in physiotherapy technique or schedule within 7 days prior to Visit 1 (Screening).
* History of lung transplantation.
* A chest radiograph at Visit 1 (Screening) or within the previous 90 days of Screening, with abnormalities indicating a significant acute finding (eg, lobar infiltrate and atelectasis, pneumothorax, or pleural effusion).
* Abnormal renal or hepatic function or serum chemistry at Visit 1 (Screening):

  * AST, ALT > 2.5 times upper limit of normal range.
  * Creatinine > 1.5 times upper limit of normal range.
* Positive pregnancy test. All women of childbearing potential will be tested.
* Female of childbearing potential who is lactating or is not practicing acceptable method of birth control (eg, hormonal or barrier methods, or IUD).
* Findings at Visit 1 (Screening) that, in the investigator's opinion, would compromise the safety of the patient or the quality of the study data.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2003-06; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 from Baseline to Day 14 | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L Gibson, Jr., MD, Principal Investigator — Children's Hospital and Regional Medica Center, Seattle, WA; George Retsch-Bogart, MD, Principal Investigator — University of North Carolina Hospitals, Chapel Hill, NC
Locations (20):
- United States (20):
  - Los Angeles, California
  - Orange, California
  - San Diego, California
  - Stanford, California
  - Denver, Colorado
  - Gainsville, Florida
  - Orlando, Florida
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Omaha, Nebraska
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Madison, Wisconsin